CLINICAL TRIAL: NCT00964444
Title: Demonstration of a New Device to Measure the Force of Delivering a Baby
Status: Completed | Type: Observational
Sponsor: Pinnacle Health System (Other)
Responsible Party: David B Peisner MD, Pinnacle Health
Other Study IDs: 6684165DP01
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Results first posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-07

CONDITIONS: Full Term Singleton Pregnancy
Keywords: Labor and delivery; Vaginal delivery

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Peisner device — The doctor/midwife stands on the device while the baby is delivered. The device measures how much force is exerted on the baby.
  Other Names: Peisner platform

SUMMARY:
This study is an observational study to prove that a new device, which measures the force of delivering a baby, (US patent 6,684,165) functions as described in the patent. This is the first time this has been used with patients.

DETAILED DESCRIPTION:
Currently, there is no way to measure how hard a doctor or midwife pulls when a baby is delivered. This device is a platform with special sensors. The doctor or midwife stands/sits on the platform while delivering the baby, and using a simple physical principle: for every action, there is an equal an opposite reaction. Prior to building the prototype and starting the study, the system and concept has been patented (US patent 6,684,165). In reality, this is not really a medical device since it does not touch the patient and does not have any effect on the delivery itself. It is merely a new type of external observation of the delivery of a baby that happens to produce useful information (the force that is exerted when the baby is delivered).

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy at term
* Singleton gestation
* Vertex presentation

Exclusion Criteria:

* Non-reassuring fetal heart rate tracing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an uncomplicated singleton pregnancy at term in active labor, who are anticipated to have a vaginal delivery.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Peisner, MD, Principal Investigator — Pinnacle Health System
Locations (1):
- Harrisburg Hospital, Harrisburg, Pennsylvania, United States

REFERENCES:
- [Derived] Peisner DB. A device that measures the pulling force and vector of delivering a baby. Am J Obstet Gynecol. 2011 Sep;205(3):221.e1-7. doi: 10.1016/j.ajog.2011.04.029. Epub 2011 Apr 24. PMID 21684515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant patients at term in early labor with a singleton vertex fetus and anticipated vaginal delivery are recruited in the labor & delivery suite of Harrisburg Hospital for this study
Pre-assignment Details: Due to the nature of the equipment, if a midwife or obstetrician was planning a bed delivery rather than using stirrups, the patient is excluded.
Groups:
- Delivery Force Study Patients: This observational study consisted of a single group of patients in active labor. The device was used to measure the force of delivering the baby. All calculations were done after the delivery was completed. Since this was an observational study, the clinical care providers did not receive the results while the patient was in the delivery suite.
Period: Overall Study
Arm/Group | Delivery Force Study Patients
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Delivery Force Study Patients
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Force Exerted on a Fetus as the Delivery Occurs
Description: The amount of force exerted on the fetus was measured in ounces. It was calculated based on measurements from the force transducers in the platform. The obstetrician stands or sits on the platform as the infant is delivered.
Time Frame: Assessment was done after the delivery
Measure: Mean (Standard Deviation); unit: ounces
Arm/Group | Delivery Force Study Patients
Number analyzed (Participants) | 10
ounces | 274.5 (107.8)

ADVERSE EVENTS:
Arm/Group | Delivery Force Study Patients
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delivery Force Study Patients (N=10)
Device failure (Pregnancy, puerperium and perinatal conditions) | 0 (0) — Since this study was observational, since the device did not affect clinical care nor touch the patient, the only potential adverse event for the study would have been device failure. The device did not fail. Therefore, there was no adverse event.

LIMITATIONS AND CAVEATS:
The trial was limited to singleton term pregnancy (37-42 weeks) patients in active labor. The study was only designed to prove that the device works and not to determine the normal range of force exerted on a fetus as it was delivered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes